CLINICAL TRIAL: NCT06368115
Title: D- PRESCRIBE-AD Phase 2(The Developing a PRogram to Educate and Sensitize Caregivers to Reduce the Inappropriate Prescription Burden in Elderly With Alzheimer's Disease Study: Trial 2)
Brief Title: A Program to Reduce Inappropriate Medications Among Older Adults With Alzheimer's Disease: Implementation Phase 2
Acronym: DPRESCRIBE-AD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Harvard Pilgrim Health Care (Other); Humana Healthcare Research, Inc. (Unknown); Carelon Research (Other)
Responsible Party: Principal Investigator, Jerry Gurwitz, Professor of Medicine, Family Medicine and Community Health, and Population & Quantitative Health Sciences, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00023453; 4R33AG069794 (NIH)
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Deprescribing; Dementia; Medication Safety
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The study design will be a prospective, randomized, "open-label" educational intervention trial with three arms: (1) a combined patient/caregiver and provider educational intervention mailed one time; (2) a combined patient/caregiver and provider educational intervention mailed two times; and (3) usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Mailing (Experimental): A combined patient/caregiver and provider educational intervention with one mailing to each.
  Interventions: Other: Educational Materials
- Two Mailings (Experimental): A combined patient/caregiver and provider educational intervention with a second identical mailing, following the first within 45 days
  Interventions: Other: Educational Materials
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Educational Materials — Educational materials on inappropriate prescribing and deprescribing.
  Arms: Single Mailing; Two Mailings

SUMMARY:
Potentially inappropriate prescribing includes the use of medications that may no longer be necessary or that may increase the risk of harm. Inappropriate prescribing can increase the overall symptom burden, and negatively affect health-related quality of life and function. The inappropriate prescription of certain drug categories such as sedative/hypnotics, antipsychotics, and strong anticholinergic agents poses particular risks for older adults, and may be more common among those with Alzheimer's disease and Alzheimer's disease- related dementias (AD/ADRD) due to a higher prevalence of multimorbidity and more frequent prescription of five or more medications. The D-PRESCRIBE-AD (Developing a PRogram to Educate and Sensitize Caregivers to Reduce the Inappropriate Prescription Burden in Elderly with Alzheimer's Disease) study will test a health plan-based intervention using the NIH Collaboratory's Distributed Research Network, which employs the Food and Drug Administration (FDA) Sentinel System infrastructure. The overarching goal of this randomized controlled trial is to assess the effect of a patient/caregiver- centered, multifaceted educational intervention on potentially inappropriate prescribing in patients with AD/ADRD. The research hypothesis is that education on inappropriate prescribing among patients/caregivers and their providers can reduce medication-related morbidity in patients with AD/ADRD and improve medication safety for this vulnerable population. The study population will include community-dwelling patients with AD/ADRD, identified based on diagnoses codes of AD/ADRD or use of a medication for Alzheimer's Disease, who have evidence of potentially inappropriate prescribing the three drug classes above. The trial will evaluate the effect of mailed educational interventions, including the effect of a second reminder mailing, designed to spur patient/caregiver-provider communication about medication safety (versus usual care) on the proportion of patients with inappropriate prescribing, the primary outcome of this study. The trial will be conducted in two large, national health plans.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Diagnosis of AD/ADRD based on a combination of AD/ADRD codes or treatment with a pharmacologic therapy used for AD (e.g., donepezil, rivastigmine, galantamine, and memantine) in the 365 days prior to or on cohort entry date.
2. Evidence of potentially inappropriate prescribing with antipsychotics, sedative-hypnotics, and strong anticholinergics within the past 3 months
3. Age ≥50 years of age as of cohort entry date
4. Continuous medical and pharmacy insurance coverage for at least the prior year

Patient Exclusion Criteria:

1. Evidence of residing in a nursing home or skilled nursing facility or receiving palliative care.
2. Incomplete/missing prescriber ID or incomplete contact information for either patient or prescribing provider.
3. On "do not contact" list

Provider Inclusion Criteria:

1. Prescribing provider associated with most recent prescribing of target drug.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11375 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Absence of Inappropriate Medication Prescription Dispensing | 9 months
  The primary outcome will be defined as absence of any dispensing of the targeted inappropriate prescription class from day 91 to day 270 during the 9 months following receipt of intervention. These 9 months are split into a 3-month black-out period followed by a six-month observation period, or days 91-270.

SECONDARY OUTCOMES:
Dose Change | 9 months
  Dose change (defined as > 50% reduction in dose of the selected inappropriate medication), assessed at the participant level using health claims data (outpatient dispensing) during days 91-270.
Polypharmacy | 9 months
  Proportion of patients with polypharmacy (defined as >5 active prescriptions for different agents) during days 91-270.
Rates of Health Care and Emergency Care Utilization | 9 months
  Rates of: emergency room visits; rates of hospitalizations; rates of non-acute institutional stays (e.g., skilled nursing facilities); and overall health care utilization (number of outpatient visits, days hospitalized, emergency department visits, and non-acute institutional days) during days 91-270.
Mortality | 9 months
  In-hospital all-cause mortality during days 91-270.
Switching within Classes | 9 months
  Switching of agents within the following targeted drug classes: sedative/ hypnotics, antipsychotics, highly anticholinergic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — UMass Chan Medical School; UMass Memorial Medical Center;
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No